CLINICAL TRIAL: NCT06279572
Title: Immune Profile of Acute Myeloid Leukemia Patients Receiving Azacitidine Plus Venetoclax Induction Chemotherapy: Opportunities for T-Cell Directed Immunotherapy
Brief Title: Immune Profile of Acute Myeloid Leukemia Patients Receiving Azacitidine Plus Venetoclax Induction Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-011624; NCI-2022-09618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-011624 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Fluid Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow and peripheral blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (blood collection, bone marrow aspirate): Patients undergo blood sample collection and bone marrow aspirate on study. Patients' medical records are reviewed.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspirate — Undergo bone marrow aspirate
  Other Names: BONE MARROW, LIQUID; Human Bone Marrow Aspirate
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study investigates the immune profile of patients receiving treatment with venetoclax plus azacitidine for acute myeloid leukemia (AML). Studying the information gathered from the immune profile from blood and bone marrow samples may help researchers understand the associated responses to the treatment of patients undergoing therapy of venetoclax plus azacitidine and create future immune based treatment approaches.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate immune profile of AML patients receiving venetoclax plus azacitidine induction chemotherapy.

SECONDARY OBJECTIVE:

I. To determine clinical responses based on immune infiltrated vs immune depleted subtypes of AML receiving azacitidine and venetoclax chemotherapy.

OUTLINE: This is an observational study.

Patients undergo blood sample collection and bone marrow aspirate on study. Patients' medical records are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 yrs of age with diagnosis of acute myeloid leukemia who received azacitidine plus venetoclax chemotherapy
* Treatment naive adult acute myeloid leukemia patients

Exclusion Criteria:

* Acute myeloid leukemia patients receiving azacitidine and venetoclax as salvage therapy will be excluded
* Patients who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myeloid leukemia who received azacitidine plus venetoclax chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune profile of treatment naive acute myeloid leukemia (AML) patients receiving azacitidine plus venetoclax chemotherapy | Baseline (at enrollment)
  Assessed using additional biospecimen samples collected during standard of care procedures (10-15 ml of peripheral blood and 10 ml of bone marrow aspirate samples). Specimens will be cryopreserved and stored for cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Talha Badar, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials